CLINICAL TRIAL: NCT00982670
Title: Association of the Metabolic Syndrome and Systemic Lupus Erythematosus in Taiwan
Brief Title: A Study of the Metabolic Syndrome in Patients With Systemic Lupus Erythematosus
Status: Completed | Type: Observational
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Chun-Chen Yang, Far Eastern Memorial Hospital
Other Study IDs: FEMH-96-D-032
Record Dates: First submitted 2009-09-22; First posted 2009-09-23 (Estimated); Last update posted 2009-09-23 (Estimated); Status verified 2009-09

CONDITIONS: Metabolic Syndrome; Cardiovascular Risk Factors; Systemic Lupus Erythematosus
Keywords: Metabolic syndrome; Systemic lupus erythematosus
MeSH Terms: conditions — Metabolic Syndrome; Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Stored serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Systemic lupus erythematosus: Patients should fulfill the diagnostic criteria of the 1997 American College of Rheumatology for systemic lupus erythematosus
- Normal control: Age- and sex-matched health volunteers will serve as controls.

SUMMARY:
An increased prevalence of the metabolic syndrome has been found in patients with systemic lupus erythematosus in recent years.

DETAILED DESCRIPTION:
This study will investigate the prevalence of the metabolic syndrome in patients with SLE in Taiwan. We expect our study will provide further understanding of the association between SLE and metabolic syndrome, which may give direction to prevent late cardiovascular morbidity and mortality in SLE patients.

ELIGIBILITY:
Inclusion Criteria:

* Persons aged 18 and above.
* Persons fulfill the diagnostic criteria of the 1997 American College of Rheumatology for systemic lupus erythematosus in the patient group.

Exclusion Criteria:

* Exclude a history myocardial infarction, angina or stroke.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Persons aged 18 and above.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2008-07; Primary Completion 2008-12 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
The prevalence of the metabolic syndrome in patients with systemic lupus erythematosus in Taiwan | One year

CONTACTS AND LOCATIONS:
Overall Officials: Chun-Chen Yang, MD, Principal Investigator — Far Eastern Memorial Hospital
Locations (1):
- Far Eastern Memorial Hospital, Pan-Chiao, Taipei, Taiwan